CLINICAL TRIAL: NCT03534362
Title: Randomized Trial of Propel Stent vs Kenalog-soaked Nasopore After Frontal Drill-out
Brief Title: Propel Stent vs Kenalog-soaked Nasopore After Frontal Drill-out
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient resources available to complete the study
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Joseph Brunworth, MD, Assistant Professor, St. Louis University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 28525
Record Dates: First submitted 2018-04-30; First posted 2018-05-23 (Actual); Results first posted 2020-04-21 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Stent; Sinusitis, Frontal
Keywords: Propel Stent; Nasopore
MeSH Terms: conditions — Frontal Sinusitis

STUDY DESIGN:
Intervention Model Description: Single-blind (Subject) randomized, active control study. Subjects will be randomized 1:1 using the rand function in Microsoft Excel program.
Who Masked: Participant
Masking Description: Patients eligible for the study and consenting to participate will be randomly assigned to one of two treatment groups: 1) Nasopore group will receive frontal drill out procedure as indicated with Kenalog-soaked Nasopore stent applied to the post-operative outflow tract and 2) Propel stent group will receive frontal drill out procedure as indicated followed by Propel stent placement applied to the post-operative outflow tract.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Nasopore Group (Active Comparator): Nasopore group will receive frontal drill out procedure as indicated with Kenalog-soaked Nasopore stent intervention applied to the post-operative outflow tract.
  Interventions: Device: Nasopore
- Propel Stent Group (Active Comparator): Propel stent group will receive frontal drill out procedure as indicated followed by Propel stent placement intervention applied to the post-operative outflow tract.
  Interventions: Device: Propel

INTERVENTIONS:
Device: Nasopore — Nasopore group will receive frontal drill out procedure as indicated with Kenalog-soaked Nasopore stent applied to the post-operative outflow tract
  Arms: Nasopore Group
Device: Propel — Propel stent group will receive frontal drill out procedure as indicated followed by Propel stent placement applied to the post-operative outflow tract.
  Arms: Propel Stent Group

SUMMARY:
Surgery on the frontal sinus is done for patients who have sinus problems that do not respond to medications. It involves making an opening within the right and left frontal sinus of the nose to help it drain. For severe frontal sinus disease, the sinus is widely opened and the left and right sinuses become one large sinus. This is done with sharp instruments and rigid endoscopes placed through the nostrils. While the sinus heals after surgery, a stent or steroids or both may be used to try to help make sure that the opening does not close back up. Two current options for this are Propel stents and steroid-soaked Nasopore. Propel stents are FDA-approved. Nasopore and Kenalog injection are both FDA-approved, but their use together is part of the study and not specifically FDA-approved. A previous study shows that Propel stents are useful to reduce scarring in other frontal sinus procedures. We would like to know whether this is true in larger frontal sinus surgery where one common cavity is made and whether both steroid-containing stents are the same.

DETAILED DESCRIPTION:
Endoscopic sinus surgery is commonly used to manage chronic inflammatory frontal sinus disease that is not adequately controlled with medical therapy alone. In recalcitrant cases, a more extensive procedure called the modified endoscopic Lothrop procedure or frontal drill-out (FDO) procedure is often performed. The frontal drill-out procedure is performed endoscopically and its goal is to create one large common cavity between the left and right frontal sinuses and nasal cavities to allow adequate drainage and communication for subsequent drug delivery through sinonasal irrigations if indicated. Failure of this procedure is most commonly the results of re-stenosis of the outflow tract due to scarring, adhesions, or progressive disease such as polyposis. One meta analysis assessing the long-term complications of frontal drillouts reported an overall failure rate to be 13.9%, defined as those individuals needing further surgery. Another clinical trial reported a failure rate for a 200-person study to be 30%.

Placing a steroid-eluding biodegradable stent into the sinonasal cavities after surgery is thought to reduce the occurrence of re-stenosis, both by physically stenting the opening and by treating resultant inflammation with corticosteroid. Propel stents are made of synthetic dissolvable polymer that contains a corticosteroid (mometasone furoate) and has been FDA-approved to stent and reduce inflammation over 30 days. Similarly, Nasopore is an FDA-approved fragmentable nasal dressing that is used as a stent. Kenalog soaking the Nasopore is thought to act as the functional equivalent of the mometasone furoate found in the Propel stent, but this use is investigational. The effect of stenting and its consequences on the outcomes of FDO specifically has also not been well studied.Recent randomized-controlled trial of Propel stent placement after frontal sinusotomy (a less extensive form of frontal sinus surgery compared to FDO procedure) showed improvement in outcomes compared to no stent placement and no major complications.There are no known randomized-controlled trials to date of propel stent placement or Nasopore-soaked Kenalog placement after FDO procedure. We wish, therefore, to perform a randomized trial to compare the efficacy and outcomes of Nasopore-soaked kenalog versus propel stenting.

ELIGIBILITY:
Inclusion Criteria:

* Patients able to speak and understand English
* Patients for whom frontal drill out procedure is medically indicated

Exclusion Criteria:

* Patients who are cognitively impaired and unable to consent
* Patients who are not candidates for Frontal Drill out
* Patients with contraindications to PROPEL Mini sinus implant or Kenalog soaked nasopore: known hypersensitivity to mometasone furoate, Kenalog, lactide, glycolide or caprolactone copolymers
* Non-English speaking patients

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-04-13 (Actual); Primary Completion 2019-09-23 (Actual); Study Completion 2019-09-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joe D Brunworth, MD, Principal Investigator — St. Louis University
Locations (1):
- Saint Louis Universtiy, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gross CW, Harrison SE. The modified Lothrop procedure: indications, results, and complications. Otolaryngol Clin North Am. 2001 Feb;34(1):133-7. doi: 10.1016/s0030-6665(05)70301-7. PMID 11344068
- [Background] Anderson P, Sindwani R. Safety and efficacy of the endoscopic modified Lothrop procedure: a systematic review and meta-analysis. Laryngoscope. 2009 Sep;119(9):1828-33. doi: 10.1002/lary.20565. PMID 19554631
- [Background] Eloy P, Vlaminck S, Jorissen M, Hellings P, Timmermans M, Daele J, Ransky P, Hassid S, Van Zele T, Bachert C, Poirrier AL, Bertrand B. Type III frontal sinusotomy: surgical technique, indications, outcomes, a multi-university retrospective study of 120 cases. B-ENT. 2011;7 Suppl 17:3-13. PMID 22338369
- [Background] Weber RK, Hosemann W. Comprehensive review on endonasal endoscopic sinus surgery. GMS Curr Top Otorhinolaryngol Head Neck Surg. 2015 Dec 22;14:Doc08. doi: 10.3205/cto000123. eCollection 2015. PMID 26770282
- [Background] Hunter B, Silva S, Youngs R, Saeed A, Varadarajan V. Long-term stenting for chronic frontal sinus disease: case series and literature review. J Laryngol Otol. 2010 Nov;124(11):1216-22. doi: 10.1017/S0022215110001052. Epub 2010 May 20. PMID 20482950
- [Background] Hoyt WH 3rd. Endoscopic stenting of nasofrontal communication in frontal sinus disease. Ear Nose Throat J. 1993 Sep;72(9):596-7. PMID 8223289
- [Background] Ting JY, Wu A, Metson R. Frontal sinus drillout (modified Lothrop procedure): long-term results in 204 patients. Laryngoscope. 2014 May;124(5):1066-70. doi: 10.1002/lary.24422. Epub 2013 Nov 13. PMID 24114727
- [Background] Huang Z, Hwang P, Sun Y, Zhou B. Steroid-eluting sinus stents for improving symptoms in chronic rhinosinusitis patients undergoing functional endoscopic sinus surgery. Cochrane Database Syst Rev. 2015 Jun 10;2015(6):CD010436. doi: 10.1002/14651858.CD010436.pub2. PMID 26068957
- [Background] Smith TL, Singh A, Luong A, Ow RA, Shotts SD, Sautter NB, Han JK, Stambaugh J, Raman A. Randomized controlled trial of a bioabsorbable steroid-releasing implant in the frontal sinus opening. Laryngoscope. 2016 Dec;126(12):2659-2664. doi: 10.1002/lary.26140. Epub 2016 Jul 1. PMID 27363723

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Because only 1 participant was recruited and enrolled, results are not reported in order to protect the confidentiality of the participant.
Groups:
- Nasopore Group: Nasopore group will receive frontal drill out procedure as indicated with Kenalog-soaked Nasopore stent intervention applied to the post-operative outflow tract.
  Nasopore: Nasopore group will receive frontal drill out procedure as indicated with Kenalog-soaked Nasopore stent applied to the post-operative outflow tract
  Because only 1 participant was recruited and enrolled, results are not reported in order to protect the confidentiality of the participant.
- Propel Stent Group: Propel stent group will receive frontal drill out procedure as indicated followed by Propel stent placement intervention applied to the post-operative outflow tract.
  Propel: Propel stent group will receive frontal drill out procedure as indicated followed by Propel stent placement applied to the post-operative outflow tract.
  Because only 1 participant was recruited and enrolled, results are not reported in order to protect the confidentiality of the participant.
Period: Overall Study
Arm/Group | Nasopore Group | Propel Stent Group
Started | 0 | 1
Completed | 0 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Only 1 subject enrolled
Groups:
- Total: Total of all reporting groups
Arm/Group | Nasopore Group | Propel Stent Group | Total
Number analyzed (Participants) | 0 | 1 | 1
Age, Categorical [Count of Participants; unit: Participants] — Because only 1 participant was recruited and enrolled, results are not reported in order to protect the confidentiality of the participant. Population: Because only 1 participant was recruited and enrolled, results are not reported in order to protect the confidentiality of the participant.
Sex: Female, Male [Count of Participants; unit: Participants] — Because only 1 participant was recruited and enrolled, results are not reported in order to protect the confidentiality of the participant. Population: Because only 1 participant was recruited and enrolled, results are not reported in order to protect the confidentiality of the participant.
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants] — Because only 1 participant was recruited and enrolled, results are not reported in order to protect the confidentiality of the participant.
  participants
    United States |  | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline of Sino-Nasla Outcome Test (SNOT-22) Scores
Description: To compare the difference in mean post-operative SNOT-22 scores between the Propel stent and Nasopore groups.
Time Frame: After the surgery, we will ask patients to follow up 5 times: post-operatively once between week 1-2, once between week 6-8, month 6, month 12, and month 24.
Population: Because only 1 participant was recruited and enrolled, results are not reported in order to protect the confidentiality of the participant.
Arm/Group | Nasopore Group | Propel Stent Group
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Surgical Postoperative Complications, Devices
Description: To compare the incidence of other surgical postoperative complications (diagnosed post-operative cerebrospinal fluid (CSF) leak, epistaxis requiring treatment, adhesions) between Propel stent and Nasopore.
Time Frame: as for outcome 1
Population: as for outcome 1
Arm/Group | Nasopore Group | Propel Stent Group
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Surgical Postoperative Complications, Frontal Sinus Pathology
Description: To ascertain the incidence of surgical complications based on the specific frontal sinus pathology.
Time Frame: as for outcome 1
Population: as for outcome 1
Arm/Group | Nasopore Group | Propel Stent Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 24 months
Description: Because only 1 participant was recruited and enrolled, results are not reported in order to protect the confidentiality of the participant.
Arm/Group | Nasopore Group | Propel Stent Group
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/1
Other Adverse Events (participants affected / at risk) | 0/0 | 0/1

LIMITATIONS AND CAVEATS:
Because only 1 participant was recruited and enrolled, results are not reported in order to protect the confidentiality of the participant.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-13): https://cdn.clinicaltrials.gov/large-docs/62/NCT03534362/Prot_SAP_000.pdf